CLINICAL TRIAL: NCT04786067
Title: Use of Donor Derived-cell Free DNA (AlloSure) to Facilitate Belatacept Monotherapy in Kidney Transplant Patients
Brief Title: Use of DNA Testing to Help Transition Kidney Transplant Recipients to Belatacept-only Immunosuppression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: CareDx (Industry)
Responsible Party: Principal Investigator, David Wojciechowski, Medical Director of the Kidney Transplantation Program, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2020-1339; CTA202012-0033 (Other Grant/Funding Number: CareDx)
Record Dates: First submitted 2021-02-23; First posted 2021-03-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-02

CONDITIONS: Kidney Transplant Immunosuppression
MeSH Terms: interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Immunosuppression Taper (Experimental): Patients included in this arm are kidney transplant recipients with stable kidney function currently on or are converting to a Belatacept based immunosuppression regimen. Eligible patients who are deemed immune quiescent after a 3 month monitoring period will undergo sequential withdrawal of immunosuppression medications over a 12 month period from a three drug regimen to a Belatacept only immunosuppression regimen. During the total 15 month period patients will be monitored with monthly clinic visits, blood draws for routine monitoring as well as donor derived cell free DNA and genetic testing through KidneyCare to monitor immune suppression.
  Interventions: Drug: Belatacept

INTERVENTIONS:
Drug: Belatacept — Patients will have tapering of their multi-drug immunosuppression, until Belatacept is the sole medication in their immunosuppression regimen. Belatacept will be administered as an infusion, as is routinely done clinically.

SUMMARY:
The purpose of the study is to identify kidney transplant patients that can be transitioned from multi-drug immunosuppression therapy to Belatacept monotherapy, using cell free DNA and gene expression as markers of immune quiescence. The primary objective will be to determine if donor derived-cell free DNA (AlloSure) can be utilized to facilitate Belatacept monotherapy, and to determine if Belatacept is safe and effective as immunosuppression in kidney transplant recipients. The secondary objective is to determine the utility of AlloMap as a predictor of immune quiescence and tolerance of immunosuppressive de-escalation to Belatacept monotherapy, and to evaluate the performance of iBox in predicting adverse outcomes in patients transitioned to Belatacept monotherapy

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years) recipients of a kidney-only transplant, including re-transplants
* Non-HLA identical Living or Deceased Donor Grafts
* Able to provide informed consent
* Absence of donor specific antigens
* Stable renal function (eGFR>40mL/min for 3 months prior to enrollment)
* Patients treated with Belatacept as part of de novo immunosuppression or converted to Belatacept with stable kidney function for 3 months (as stated above)
* Patients who underwent kidney transplantation at least 9 months prior to study entry

Exclusion Criteria:

* Prior or concurrent non-kidney organ transplants
* Presence of BK nephropathy in current graft
* Recipient on any other investigational drug in the 12 weeks prior to inclusion
* Patient with history of recent (<3mo), recurrent, or severe (Banff Grade 2 or greater or unable to be treated with steroids) acute rejection episodes
* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial
* Significant hepatic impairment
* Bilateral kidney transplantation
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with acute kidney graft rejection | 12 months after the date of the first immunosuppression taper
  Number of patients with Acute kidney graft rejection confirmed by biopsy by 2017 Banff Criteria.
  Incidence of biopsy proven acute kidney graft rejection at 12 months after the start of immunosuppression taper

SECONDARY OUTCOMES:
Number of patients who died | 12 months after the start of immunosuppression wean, up to 36 months
  Incidence of death will be measured from 12 months after the start of immunosuppresion wean, up to 36 months
Number of patients with kidney graft failure | 12 months after the start of immunosuppression wean
  Incidence of kidney graft failure will be measured from the start of immunosuppresion wean until 12 months after. Graft failure is defined as date of patient death or date of retransplant
Mean change in Estimated Glomerular Filtration Rate (eGFR) | Baseline, 12 months after the start of immunosuppression wean
  Estimated glomerular filtration rate (eGFR) in blood will be measured at the beginning of enrollment and the difference will be measured to the end of the study as a measure of change in kidney function.
Number of participants with Proteinuria | 12 months after the start of immunosuppression wean
  Proteinuria will be detected by a semiquantitative method of the protein concentration in urine.
Number of participants with appearance of de-novo donor specific antibodies (dnDSA) | 12 months after the start of immunosuppression wean
  HLA type I and type II in blood will be used to detect the presence of de-novo donor specific antibodies (dnDSA)
Negative predictable value as measured by AlloMap® | 12 months after the start of immunosuppression wean
  Negative predictable value measured by AlloMap®, expressed as a percent, that the patient is not experiencing rejection at the time of testing.
  AlloMap® is a panel of 20 gene assays, 11 informative and 9 used for normalization and/or quality control, which produces gene expression data used in the calculation of an AlloMap test score - an integer ranging from 0 to 40. Compared with patients in the same post- transplant period, the lower the score, the lower the probability of acute cellular rejection at the time of testing.
Mean prediction score of allograft loss as measured by iBox | 12 months after the start of immunosuppression wean
  iBox is the validated tool for predicting the risk of kidney transplant loss based on artificial intelligence. Range of score is 0%-100%, higher score indicates better kidney survival.

CONTACTS AND LOCATIONS:
Overall Officials: David Wojciechowski, DO, Principal Investigator — University of Texas Southwestern Medical Center; Cyrus Feizpour, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No